CLINICAL TRIAL: NCT05026372
Title: Two-Session Couples Class to Improve Relationship Health
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Participant drop out exceeded expectations (out of 63 couples randomized, 18 completed follow up). Study may be resumed with revised procedures for preventing drop out.
Sponsor: Sam Houston State University (Other)
Responsible Party: Principal Investigator, Chelsea Ratcliff, Assistant Professor, Sam Houston State University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB-2019-123
Record Dates: First submitted 2021-08-23; First posted 2021-08-30 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-04

CONDITIONS: Stress
Keywords: couples stress, health, psychology

STUDY DESIGN:
Intervention Model Description: The intervention conditions are divided into Mindfulness + Compassion (MC), Mindfulness + Gratitude (MG), Mindfulness + Value-Based Living (MV), and Attention Control (AC)) on Mindfulness (FFMQ).
Who Masked: Participant
Masking Description: Participants will not be informed of their group condition, i.e., MC, MG, MV, or AC.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Mindfulness + Compassion (MC) (Experimental): For participants randomized to the MC condition will focus on compassion and creating positive emotions. This session will include techniques such as guided visualizations and a loving kindness meditation that are intended to facilitate connection with their partners. During this session, couples will also learn the ground rules of mindful and compassionate listening and sharing, as they will be asked to engage in an emotional disclosure task. The instructor will go over the homework assignment. The interventionist will review the tools the couples had learned over the course of this program and help them proactively identify strategies to continue to implement them into their lives. Couples will receive instructions on how to continue with this program when no longer meeting with the interventionist.
  Interventions: Behavioral: Mindfulness Compassion (MC)
- Mindfulness + Gratitude (MG) (Experimental): Session 2 for participants randomized to group MG will focus on gratitude. Participants will be taught to reflect on things, events, and people which they are grateful for via a gratitude meditation. Couples will share their experiences of practicing gratitude. The instructor will remind the couple of ground rules prior to the emotional disclosure exercise and facilitate if necessary during the sharing. Each member of the couple will take turn in sharing with and listening to their partner. The instructor will go over the homework assignment. The interventionist will review the tools the couples had learned over the course of this program and help them proactively identify strategies to continue to implement them into their lives. Couples will receive instructions on how to continue with this program when no longer meeting with the interventionist.
  Interventions: Behavioral: Mindfulness Gratitude (MG)
- Mindfulness + Value-Based Living (MV) (Experimental): Session 2 for participants randomized to group MV will focus on learning strategies to live life according to their values. They will first engage in a reflection exercise to help identify their values, and then complete a worksheet. Couples will brain storm together strategies to ensure that their lives reflect their self-identified values. The instructor will go over the homework assignment. The interventionist will review the tools the couples had learned over the course of this program and help them proactively identify strategies to continue to implement them into their lives. Couples will receive instructions on how to continue with this program when no longer meeting with the interventionist.
  Interventions: Behavioral: Mindfulness Value-Based Living (MV)
- Attention Control (AC) (No Intervention): For participants randomized to the AC condition, both sessions will focus on discussing issues and themes that emerge for couples, such as communication and perceived supportiveness. Utilizing a reflective listening approach, the interventionist will focus on encouraging participants to share concerns related to their daily experiences. Unlike in the MC, MG, and MV groups, the interventionist will not offer advice, support (other than reflective listening) or any other tools to participants. Additionally, the interventionist will not probe for deep emotional disclosure. Please see the appendix for the session outline. We believe a control group that discusses daily relationship-related concerns serves as an excellent comparison condition in this study since it is viewed as credible by participants and equates for time and attention as well as nonspecific treatment effects such as those provided through social interactions.

INTERVENTIONS:
Behavioral: Mindfulness Compassion (MC) — The interventionist will review the tools the couples had learned over the course of this program and help them proactively identify strategies to continue to implement them into their lives. Couples will receive instructions on how to continue with this program when no longer meeting with the interventionist.
  Arms: Mindfulness + Compassion (MC)
Behavioral: Mindfulness Gratitude (MG) — The interventionist will review the tools the couples had learned over the course of this program and help them proactively identify strategies to continue to implement them into their lives. Couples will receive instructions on how to continue with this program when no longer meeting with the interventionist.
  Arms: Mindfulness + Gratitude (MG)
Behavioral: Mindfulness Value-Based Living (MV) — The interventionist will review the tools the couples had learned over the course of this program and help them proactively identify strategies to continue to implement them into their lives. Couples will receive instructions on how to continue with this program when no longer meeting with the interventionist.
  Arms: Mindfulness + Value-Based Living (MV)

SUMMARY:
This study will compare the effect of three different stress reduction intervention techniques compared to a non-intervention control group on the psychological and relationship functioning in 40 romantic couples. The current study will serve two purposes. Results will inform future efforts to develop effective brief stress reduction interventions for physically healthy couples and will inform future iterations of stress reduction-based intervention for cancer patients and their caregivers.

The investigators hypothesize that couples in the three stress-reduction interventions will report greater relationship health and greater mindfulness after the intervention than couples in the non-intervention control group. The investigators also hypothesize that the stress-reduction groups will be most beneficial for individuals who report higher distress, indifferent relationship style, and insecure attachment at baseline.

DETAILED DESCRIPTION:
Participants will be randomly assigned to one of four conditions, each of which involve participating in two 45-minute sessions (via Zoom) with a study interventionist. Sam Houston State University (SHSU) clinical psychology master's or doctoral students or graduates of the SHSU clinical psychology master's program will implement the mind-body intervention, under the supervision of Dr. Chelsea Ratcliff, who is a licensed psychologist. Dr. Ratcliff will provide weekly group supervision to all students implementing the treatment.

Participation in this study will last a total of 6 weeks (+/- 1 week). The T1 survey will last approximately 45 minutes. Within 1 week of both partners completing baseline, eligible dyads will be scheduled for Session 1. For the intervention, all participants will be emailed a PDF of the appropriate workbook prior to Session 1. Participants will also be informed that they may pick up a hard copy (printed version).

For participants in the stress-reduction groups, after each session the interventionist will send each participant an email with: 1) the audio recording of the appropriate guided stress-reduction activity (transcript provided in workbook), 2) a fillable PDF document with instructions regarding completing and documenting home-practice, and 3) a link to a Qualtrics survey that asks them to evaluate their experience in the session. The instructor will also inform participants that they may pick up hard copies of all session materials if it is convenient/preferable. For participants in the non-intervention control group, the interventionist will email each participant a link to a Qualtrics survey that asks them to evaluate their experience in the session.

Session 2 will take place approximately 1 week after Session 1. After completing session 2, the interventionist will send a link to another Qualtrics survey that asks them to evaluate their experience in the session.

Within 1 week of completing Session 2, both members of the dyad will be emailed the link to the second Qualtrics survey (T2), which will last approximately 30 minutes. Finally, within 1 month (+/- 1 week) of completing Session 2, both members of the dyad will be emailed the third Qualtrics survey (T3), which will last approximately 20 minutes.

ELIGIBILITY:
Inclusion Criteria:

ADULT ROMANTIC COUPLES in a relationship for a minimum of 6 months COHABITATING for a minimum of 6 months STRESS. At least one member of the romantic dyad reports stress above the normative mean for young adults (i.e., Perceived Stress Scale score > 17; Cohen & Janicki-Deverts, 2012).

Exclusion Criteria:

INDIVIDUALS UNDER AGE 18: This study only involves adult participants. NON-ENGLISH SPEAKING INDIVIDUALS: This study only involves participants who can speak English.

ATTENDING PSYCHOTHERAPY: This stud only involves individuals who are not currently (self-defined) participating in psychotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2019-05-29 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Perceived Stress Scale | Within 1 week of treatment ending
  Perceived Stress Scale (PSS) (Cohen & Janicki-Deverts, 2012) is a 10-item scale to measure stress. Scores range from 0-40, with higher scores indicating greater perceived stress
Perceived Stress Scale | 1 month after treatment ends
  Perceived Stress Scale (PSS) (Cohen & Janicki-Deverts, 2012) is a 10-item scale to measure stress. Scores range from 0-40, with higher scores indicating greater perceived stress

SECONDARY OUTCOMES:
Dyadic Adjustment Scale Total Score | within 1 week of treatment ending
  Dyadic Adjustment Scale (DAS-7) (Hunsley, Best, Lefebvre, & Vito, 2001; Spanier, 1976) is a 7-item scale designed to measure adjustment and satisfaction among married or cohabitating couples. Scores range from 0 to 36, with a higher score indicating more positive relationship quality. It has been used in sample of college-aged couples in previous literature.
Dyadic Adjustment Scale Total Score | 1 month after treatment ends
  Dyadic Adjustment Scale (DAS-7) (Hunsley, Best, Lefebvre, & Vito, 2001; Spanier, 1976) is a 7-item scale designed to measure adjustment and satisfaction among married or cohabitating couples. Scores range from 0 to 36, with a higher score indicating more positive relationship quality. It has been used in sample of college-aged couples in previous literature.
Five Facet Mindfulness Scale Total Score | Within 1 week of treatment completion
  Five Facet Mindfulness Scale (FFMQ) (Baer, Smith, Hopkins, Krietemeyer, & Toney, 2006) is a 39-item scale based on a factor analytic study of five independently developed mindfulness questionnaires, which yielded five factors of mindfulness: observing, describing, acting with awareness, non-judging of inner experience, and non-reactivity to inner experience. Total scores range from 39-196 with higher scores indicating greater trait mindfulness.
Five Facet Mindfulness Scale Total Score | 1 month after treatment ends
  Five Facet Mindfulness Scale (FFMQ) (Baer, Smith, Hopkins, Krietemeyer, & Toney, 2006) is a 39-item scale based on a factor analytic study of five independently developed mindfulness questionnaires, which yielded five factors of mindfulness: observing, describing, acting with awareness, non-judging of inner experience, and non-reactivity to inner experience. Total scores range from 39-196 with higher scores indicating greater trait mindfulness.

OTHER OUTCOMES:
Acceptance & Action Questionnaire-II Total Score | Within 1 week of treatment completion
  Acceptance & Action Questionnaire-II (AAQ-II), a 10 question measure of psychological flexibility (Bond et al., 2011). Scores range from 20-70, with higher scores representing greater psychological flexibility.
Acceptance & Action Questionnaire-II Total Score | 1 month after treatment ends
  Acceptance & Action Questionnaire-II (AAQ-II), a 10 question measure of psychological flexibility (Bond et al., 2011). Scores range from 20-70, with higher scores representing greater psychological flexibility.
Center for Epidemiologic Studies Depression Scale | Within 1 week of treatment completion
  Center for Epidemiologic Studies Depression Scale (CES-D; Radloff, 1977) a 20-item self-report measure of depression. Scores range from 0-60 with higher scores indicating greater depression symptoms.
Center for Epidemiologic Studies Depression Scale | 1 month after treatment ends
  Center for Epidemiologic Studies Depression Scale (CES-D; Radloff, 1977) a 20-item self-report measure of depression. Scores range from 0-60 with higher scores indicating greater depression symptoms.
Medical Outcomes Study 36-item Short-Form Survey (SF-36) Physical Component Summary (PCS) | Within 1 week of treatment completion
  Physical health-related QOL will be assessed with the Medical Outcomes Study 36-item short-form survey (SF-36) Physical Component Summary (Ware, Johnston, Davies-Avery, & al, 1994). Scores range from 0-100, with higher scores indicating better physical health-related QOL.
Medical Outcomes Study 36-item Short-Form Survey (SF-36) Physical Component Summary (PCS) | 1 month after treatment ends
  Physical health-related QOL will be assessed with the Medical Outcomes Study 36-item short-form survey (SF-36) physical component summary.(Ware, Johnston, Davies-Avery, & al, 1994). Scores range from 0-100, with higher scores indicating better physical health-related QOL.
Medical Outcomes Study 36-item Short-Form Survey (SF-36) Mental Component Summary (MCS) | Within 1 week of treatment completion
  Mental health-related QOL will be assessed with the Medical Outcomes Study 36-item short-form survey (SF-36) mental component summary.(Ware, Johnston, Davies-Avery, & al, 1994). Scores range from 0-100, with higher scores indicating better mental health-related QOL.
Medical Outcomes Study 36-item Short-Form Survey (SF-36) Mental Component Summary (MCS) | 1 month after treatment ends
  Mental health-related QOL will be assessed with the Medical Outcomes Study 36-item short-form survey (SF-36) mental component summary.(Ware, Johnston, Davies-Avery, & al, 1994). Scores range from 0-100, with higher scores indicating better mental health-related QOL.

CONTACTS AND LOCATIONS:
Overall Officials: Chelsea G Ratcliff, Ph.D., Principal Investigator — Sam Houston State University
Locations (1):
- Sam Houston State University, Huntsville, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided